CLINICAL TRIAL: NCT06975566
Title: Long-term Effects of Radial Artery Cannulation on Vessel Diameter, Blood Flow and Fine Motor Skills
Status: Completed | Type: Observational
Sponsor: Kartal City Hospital (Other)
Responsible Party: Principal Investigator, AKIN BİLİR, anesthesiology and reanimation specialist, intensive care subspecialist, Kartal City Hospital
Other Study IDs: radial artery study
Record Dates: First submitted 2025-05-01; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Radial Artery; Ultrasound; Fine Motor Skills
Keywords: Catheterization; Regional blood flow; Fine motor skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: radial artery catheterization

SUMMARY:
The present study aims to investigate hemodynamic changes in radial and ulnar artery blood flow following radial artery cannulation performed in elective surgical cases under operating room conditions using Doppler ultrasonography. Additionally, it aims to evaluate the long-term impact of this procedure on vascular flow parameters and fine motor function.

DETAILED DESCRIPTION:
This prospective self controlled study included 50 patients aged 18-80 years with an ASA physical status of 1-3 who required arterial cannulation for planned surgical procedures in the cardiovascular surgery operating rooms of Pamukkale University Faculty of Medicine. Before the procedure, radial and ulnar artery Doppler parameters (peak systolic velocity, end-diastolic velocity, resistance index, pulsatility index, and mean volume flow) were measured for all patients, along with Purdue Pegboard scores for fine motor skill assessment. Post-cannulation Doppler parameters were evaluated at seven different time points over three months, while fine motor skill scores were measured twice more during follow-up.

ELIGIBILITY:
Inclusion Criteria:

indication for radial artery cannulation

Exclusion Criteria:

emergency surgery inadequate collateral blood flow

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing surgical intervention at Pamukkale University Faculty of Medicine, Department of Cardiovascular Surgery, between June and September 2016. Patients aged 18 to 80 years, scheduled for elective surgery, and with an indication for radial artery cannulation were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
90 DAY FOLLOW-UP PERIOD | From the first measurement before cannulation to the last measurement after 90 days
  Fifty patients requiring arterial cannulation were included in this study. Before the procedure, radial and ulnar artery Doppler parameters (peak systolic velocity, end-diastolic velocity, resistance index, pulsatility index, and mean volume flow) were measured for all patients, along with Purdue Pegboard scores for fine motor skill assessment. Post-cannulation Doppler parameters were assessed at seven different time points over three months, while fine motor skill scores were measured twice more.
90 DAY FOLLOW-UP PERIOD | From the first measurement before cannulation to the last measurement after 90 days
  Fifty patients requiring arterial cannulation were included in this study. Purdue Pegboard scores were measured for fine motor skill assessment of all patients before the procedure. Over three months fine motor skill scores were measured twice more.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Desrosiers J, Hebert R, Bravo G, Rochette A. Age-related changes in upper extremity performance of elderly people: a longitudinal study. Exp Gerontol. 1999 Jun;34(3):393-405. doi: 10.1016/s0531-5565(99)00018-2. PMID 10433393
- [Background] Taneja K, Jain R, Sawhney S, Rajani M. Occlusive arterial disease of the upper extremity: colour Doppler as a screening technique and for assessment of distal circulation. Australas Radiol. 1996 Aug;40(3):226-9. doi: 10.1111/j.1440-1673.1996.tb00391.x. PMID 8826723
- [Background] Numaguchi A, Adachi YU, Aoki Y, Ishii Y, Suzuki K, Obata Y, Sato S, Nishiwaki K, Matsuda N. Radial artery cannulation decreases the distal arterial blood flow measured by power Doppler ultrasound. J Clin Monit Comput. 2015 Oct;29(5):653-7. doi: 10.1007/s10877-014-9648-5. Epub 2014 Dec 16. PMID 25516161